CLINICAL TRIAL: NCT02358278
Title: Evaluation and Implementation of the "Paediatric Anesthesia Emergence Delirium Scale" (PAED) in the PACU in Children Under 14 Years of Age
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Camus Virchow -Klinikum, Charite University, Berlin, Germany
Other Study IDs: EI-PAED
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Paediatric Anesthesia Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to determine the incidence and characteristics of Emergence Delirium (ED) in children aged 0 - 13 undergoing general anesthesia and being taken care of at the paediatric PACU of the Charité Campus Virchow-Clinic. Therefore the "Paediatric Anesthesia Emergence Delirium Scale" (PAED) is used. In order to measure the patient's pain level, age-appropriate pain scales (CHIPPS or FPS-R) are applied. Risk factors for the occurrence of ED are to be determined and therapeutic approaches in case of an occurring ED are to be evaluated. Finally the future implementation of ED-monitoring in the PACU is to be prepared.

DETAILED DESCRIPTION:
Emergence Delirium is a widely known phenomenon during the recovery phase after general anesthesia in children. In spite of the existence of a vast number of studies dealing with this topic and even after the development of a validated measurement tool for ED (PAED-Scale, Sikich et al. 2004), data regarding incidence, risk factors and treatment of ED vary considerably.

This study seeks to determine the actual incidence and characteristics of Emergence Delirium (ED) in children at the paediatric PACU of the Charité Campus Virchow-Clinic. Therefore the PAED-Scale is applied in a large population of children aged 0 - 13 years undergoing general anesthesia. In addition a clinical evaluation regarding the presence of ED is conducted by the PACU nurses on the basis of their clinical experience.

In order to preserve the possibility of minimizing the influence of postoperative pain, which has been identified as a confounding variable in the measurement of ED, an age-appropriate pain score is measured simultaneously with each PAED-Score. The Children's and Infants Postoperative Pain Scale (CHIPPS) (Büttner, 1998) is used for children aged 0 - 4 years. The Faces Pain Scale-Revised (FPS-R) (Hicks et al. 2001) is used for older children.

Besides the study aims to identify possible factors that are associated with a higher incidence of ED. Therefore perioperative data (anesthetic and analgetic agents, duration of anesthesia, premedication, volume therapy etc.) is obtained.

In case of the occurrence of ED additional data (duration of ED, treatment of ED) is collected.

All data is collected by using a questionnaire that is completed by the anesthesists and the PACU staff.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing anesthesia and being taken care of at the paediatric PACU
* Aged 0 - 13 years

Exclusion Criteria:

• None

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children (age 0-13) receiving anesthetic care for operative procedures and are cared for in the post-anesthesia care unit are monitored for emergence delirium and therapeutic measures.
Sampling Method: Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Paediatric Anesthesia Emergence Delirium (PAED) Score | It is measured until the end of post-anesthesia care unit (PACU) stay - or for a maximum of 24 hours
  (PAED) Score at four different points of time:
  1. 5 - 10 minutes after awakening
  2. At clinical signs of ED (only if applicable)
  3. After ED therapy (only if applicable)
  4. At discharge from the PACU
  Age-appropriate pain score simultaneously with each PAED Score
  * Age 0 - 4: Children's and Infants Postoperative Pain Scale (CHIPPS)
  * Age 5 - 13: Faces Pain Scale-Revised (FPS-R)

SECONDARY OUTCOMES:
Operation procedure | At time of surgery
  Kind of surgical procedure
Duration of anesthesia | At time of surgery
Induction of anesthesia (anesthetic agents) | At time of surgery
Maintenance of anesthesia (anesthetic agents) | At time of surgery
Analgesic agents | It is measured until the end of post-anesthesia care unit (PACU) stay - or for a maximum of 24 hours
Fluid balance | At time of surgery
  Fluid and volume administration and balance
Blood transfusions | They are measured until the end of PACU stay - or for a maximum of 5 days
Duration of stay in the PACU | Period of PACU stay
Duration of Emergence Delirium | It is measured until the end of PACU stay - or for a maximum of 5 days
Pharmacological treatment of Emergence Delirium | It is measured until the end of post-anesthesia care unit (PACU) stay - or for a maximum of 24 hours
Non-pharmacological treatment of Emergence Delirium | It is measured until the end of post-anesthesia care unit (PACU) stay - or for a maximum of 24 hours
Pain scores | It is measured until the end of post-anesthesia care unit (PACU) stay - or for a maximum of 24 hours
  Age 0 - 4: Children's and Infants Postoperative Pain Scale (CHIPPS)
  ◦Age 5 - 13: Faces Pain Scale-Revised (FPS-R)
Anesthesia | At time of surgery
  General Anesthesia or general anesthesia combined with regional anesthesia

OTHER OUTCOMES:
Gender | At the beginning of the investigation
Age | At the beginning of the investigation
Height | At the beginning of the investigation
Weight | At the beginning of the investigation
ASA-Classification | At the beginning of the investigation
Admission diagnosis | At the beginning of the investigation
Comorbidities | At the beginning of the investigation
Long-term medication | At the beginning of the investigation
Premedication | At the beginning of the investigation
PONV prophylaxis | At the beginning of the investigation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum (CVK) and Campus Charite Mitte (CCM), Charite - Universitätsmedizin Berlin, Berlin, Germany